CLINICAL TRIAL: NCT06437054
Title: Verification of the Efficacy/Safety of the Mixed Drug Injectable Delivery Vehicle for Treating Intractable Hearing Loss (Pilot Study)
Brief Title: Verification of the Efficacy/Safety of the Mixed Drug Injectable Delivery Vehicle for Treating Intractable Hearing Loss
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITV-2309-098-1469
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-05

CONDITIONS: Hearing Loss, Sensorineural; Hearing Loss, Sudden; Intratympanic Injection
Keywords: drug delivery; Dexamethasone; Hyaluronic acid
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Sudden | interventions — Dexamethasone; Hyaluronic Acid; Indocyanine Green

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone+Saline+ICG (Active Comparator): The experimental group received a single injection of Dexamethasone (5mg/ml) and Saline (D+Saline) mixed in a 1:1 ratio (with a possibility of a second injection if necessary). Additionally, two drops of Indocyanine Green (ICG: 25mg) were added, approximately 100μl (2.5mg/ml).
  Interventions: Drug: Dexamethasone; Other: Indocyanine green(ICG)
- Dexamethasone+Hyaluronic Acid+ICG (Experimental): The experimental group received a single injection of Dexamethasone (5mg/ml) and Hyaluronic acid (D+HA) mixed in a 1:1 ratio (with a possibility of a second injection if necessary). Additionally, two drops of Indocyanine Green (ICG: 25mg) were added, approximately 100μl (2.5mg/ml).
  Interventions: Drug: Dexamethasone; Drug: Hyaluronic acid; Other: Indocyanine green(ICG)

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 5mg/ml
  Other Names: Dexamethasone Inj (Dexamethasone disodium phosphate 5㎎) [Daewon Pharm]
Drug: Hyaluronic acid — Hyaluronic Acid 20mg/2ml
  Other Names: Hyruan Plus Inj (Sodium Hyaluronate 10.0mg) [LG Chem]
  Arms: Dexamethasone+Hyaluronic Acid+ICG
Other: Indocyanine green(ICG) — ICG 25mg
  Other Names: Cellbiongreen Inj (IndocyanineGreen 25mg) [Cellbion]

SUMMARY:
This study is a prospective, randomized pilot study. To verify an efficacy/safety of the mixed drug injectable delivery vehicle for treating intractable hearing loss. Hearing test, endoscopy of tympanic membrane and CT scans will be conducted after intratympanic treatment for evaluation.

DETAILED DESCRIPTION:
The goal of this clinical trial (pilot study) is to evaluate the Efficacy and Safety of Combined Hyaluronic Acid and Dexamethasone Treatment in Patients with Hearing Loss. The main questions it aims to answer are: • Q1. Verification of safety, • Q2. Therapeutic effect of drug injection on sensorineural hearing loss. Participants will undergo several assessment tests (Verification of adverse effects in the external and middle ear through endoscopy, Confirmation of adverse effects through imaging, Hearing test to check for additional hearing loss, Check if subjective ear fullness persists for more than a week aside from the drug effect). If there is a comparison group: Researchers will compare dexamethasone and hyaluronic acid to verify hearing improvement and safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sudden hearing loss, Meniere's disease, ototoxic hearing loss, and noise-induced hearing loss of 25dB HL at the frequency at which hearing loss occurs as a result of pure tone hearing test
* Patients whose original hearing ability has not been restored with existing standard treatment (oral, intravenous steroids)
* Those who have not participated in clinical trials within 3 months are selected as subjects

Exclusion Criteria:

* Pregnant or lactating women
* When accompanied by lesion, infection, or anatomical deformity of the outer ear, middle ear, or inner ear
* Those with liver disease or metabolic disease or a history thereof
* History of hypersensitivity to indocyanine green or iodine hypersensitivity
* History of ear surgery
* Cases with posterior labyrinth lesions
* Patients with a history of hypersensitivity to the ingredients of this drug
* In addition, serious diseases such as end-stage renal disease, end-stage liver disease, cardiovascular surgery, progressive brain tumor, progressive hemorrhage, and progressive cerebral hemorrhage are included Cases with brain disease and cancer are excluded from the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Analysis of Side Effect Rate through tympanic membrane endoscopy Imaging in 26 participants | 0, 1day and 1 week after intratympanic injection
  Confirming healing time of perforation and inflammation (Safety)
Analysis of Drug Duration through CT Imaging in 26 participants | 0, 1day and 1 week after intratympanic injection
  Checking a time duration of drug in middle and inner ear (Durability)
Comparison of Auditory Threshold Values Between Two Groups to Confirm Treatment Efficacy in 26 participants | 0, 1day, 1 week and/or 1 month after intratympanic injection
  Verifying therapeutic effect of intratympanic drug delivery vehicle (Efficacy)

IPD SHARING:
Plan to Share IPD: No